CLINICAL TRIAL: NCT02575664
Title: Effects of Low Dose Buprenorphine on Recovery After Hip or Knee Arthroplasty
Acronym: lonkkalaasta
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Collaborators: University of Eastern Finland (Other)
Responsible Party: Principal Investigator, Merja Kokki, MD, PhD, Kuopio University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KUH2011-000692-14
Record Dates: First submitted 2015-10-09; First posted 2015-10-15 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Pain; Osteoarthritis
Keywords: Pain; Arthroplasty; Buprenorphine
MeSH Terms: conditions — Pain; Osteoarthritis | interventions — Buprenorphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Buprenorphine (Experimental): Buprenorphine 5 microg/h/7days patch
  Interventions: Drug: Buprenorphine
- Placebo (Placebo Comparator): Placebo patch
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Buprenorphine — Buprenorphine 5 microg/h/7 days
  Arms: Buprenorphine
Drug: Placebo — Placebo patch
  Arms: Placebo

SUMMARY:
Buprenorphine is a highly lipophilic thebaine derivative that appears to have high affinity for mu-, kappa-, and delta-opioid receptors and low affinity for opioid receptors like 1 -receptors. It acts as a partial agonist at the mu-opioid and as a partial agonist/antagonist at the kappa-opioid, and as an antagonist at the delta opioid receptors. Buprenorphine has up to two-fold duration of action and it is approximately 30-fold more potent when compared to morphine.

Pain is a common problem in patients coming to joint arthroplastic surgery. Buprenorphine low dose patches are recommended for treatment of moderate pain for example osteoarthritis pain. It is known that well treated pain even preoperatively may prevent prolonged postsurgical pain.

In the present study the effects of low dose buprenorphine on postoperative pain and recovery were assessed.

ELIGIBILITY:
Inclusion Criteria:

* no pregnancy/lactation, reliable contraception before menopause
* elective knee or hip arthroplasty surgery
* BMI (=body mass index) 18-35 kg/m2
* obtained informed consent

Exclusion Criteria:

* buprenorphine medication
* allergy to study drugs• ikä < 18 tai >75 years

  * BMI <18 tai>35 kg/m2
  * weight below 50 kg
  * Other contraindication for the study drug

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2012-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Pain relief | time from drug patch administration up to five weeks
  Brief pain inventory
Prolonged pain after arthroplastic surgery | from time from drug patch administration up to one year
  Brief pain inventory

CONTACTS AND LOCATIONS:
Overall Officials: Merja Kokki, MD, PhD, Principal Investigator — Kuopio University Hospital
Locations (1):
- Kuopio University Hospital, Kuopio, Northern Savonia, Finland